CLINICAL TRIAL: NCT05100394
Title: Effectiveness of High Power Laser Therapy on Pain and Isokinetic Power in Athletes With Proximal Hamstring Tendinopathy: a Randomized Controlled Trial
Brief Title: Effectiveness of Laser Therapy on Proximal Hamstring Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2021-07
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Tendinopathy; Lasers
Keywords: Proximal hamstring tendinopathy; laser therapy; Pain; Muscle power
MeSH Terms: conditions — Tendinopathy; Pain | interventions — Laser Therapy; High-Energy Shock Waves; Exercise

STUDY DESIGN:
Intervention Model Description: Two-arm parallel-groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor was unaware of allocation into experimental or control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): High Power laser therapy was provided.
  Interventions: Radiation: Laser Therapy
- Control Group (Active Comparator): Conventional physiotherapy was applied including moist heat packs, US, and eccentric hamstring exercises.
  Interventions: Other: Ultrasound + Moist Heat pack + Exercises

INTERVENTIONS:
Radiation: Laser Therapy — Therapeutic laser therapy was applied.
  Arms: Experimental Group
Other: Ultrasound + Moist Heat pack + Exercises — Ultrasound therapy, a moist heat pack, and a home exercise program were given.
  Arms: Control Group

SUMMARY:
Proximal hamstring tendinopathy (PHT) is tendinopathy of the semimembranosus and/or biceps femoris/semitendinosus complex. Previous studies have shown the efficacy of laser therapy in the treatment of tendinopathy. To the best of the investigator's knowledge, no study has compared the effects of high-power LASER therapy with conventional physiotherapy programs in proximal hamstring tendinopathy patients. Therefore, this study aimed to assess the effects of high-power laser therapy on pain and muscle power in proximal hamstring tendinopathy patients.

DETAILED DESCRIPTION:
2 arms comparative pretest-posttest experimental research design with random allocation of subjects into groups (experimental and control group) using the lottery method. A total of thirty-six participants aged between 18-35 (mean age) years, were recruited in the present study. The selected participants were randomly allocated into experimental and control groups using the lottery method and website randomization.com with eighteen participants in each group. The participants and outcome assessor were kept blinded to the allocation. In the experimental group, the high-power laser was given whereas in the control group conventional physiotherapy treatment was given for 4 weeks. Conventional physiotherapy treatment included the US, moist heat pack, and home exercises. Home exercises include nordic hamstring exercises - 2 sets of 5 repetitions, 3 days/week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Athletes
* pain located deep in the buttock/posterior thigh region
* tenderness of ischial tuberosity
* hamstring muscle tightness.

Exclusion Criteria:

* Recent trauma to the posterior thigh
* Musculoskeletal disorder of ipsilateral lower extremity
* taking pain medication daily
* hypertension, malignancy, autoimmune disease, phlebitis, blood disorder.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 3 weeks.
  On a scale of 0-10, patients rate their current pain level. Higher scores mean worse outcome.
Isokinetic peak torque | 3 weeks.
  Isokinetic muscle power was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No